CLINICAL TRIAL: NCT05110222
Title: Evaluation of Cataract Lens Hardness Based on Phacoemulsificator Tip Resistance
Brief Title: Cataract Lens Hardness Based on Phaco Tip Resistance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Sponsor
Other Study IDs: 1/2021
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-09

CONDITIONS: Cataract Senile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Phacoemulsificaton tip elongation depends upon voltage once resonant frequency of piezoelectric crystals has been reached.

Purpose of the study is to record voltage data of 20 consecutive cataract surgeries in order to evaluate correlation between voltage and LOCS classification of lens nuclei using a system that deploys a feedback mechanism capable of keeping invariant elongation regardless of enountered resistence

DETAILED DESCRIPTION:
The R-Evolution (Optikon 2000 Rome, Italy) phaco machine is equipped with a patented system named "minimal stress" that used the direct piezoelectric effect from the resonant ceramics that drive the phacoemulsificator tip to assess in real time and adjust phaco tip elongation that continuously varies according to encountered resistance.

After priming in balanced salt solution, phaco tip elongation and the amount of potential difference (voltage) needed to obtain a ginev elongation in balanced solution is assessed. Once the phaco tip is used during surgery, the resistence offered by the crystalline lens material to the phaco tip reduces actual elongaton which in turn reduces the voltage produced by the directo piezometric effect. The machine uses voltage produced by actual elongation to adjust the diving voltage and therefore can ensure accurate pahco tip elongation under any condition of lens material resistance.

Purpose of the study is to record driving voltage and its variations and evaluate if there is a correlation between phaco tip resistence and drving voltage.

This is evaluated both in vitro activating the phaco tip in increasingly dense glycerol solutions and in real life phaco surgery recording the voltage requested by phaco tip resistence and correlating it to the classification of lens opacity (LOCS III system) clinically used to grade cataract hardness.

ELIGIBILITY:
Inclusion Criteria: diagnosis of nuclear or cortical cataract

Exclusion Criteria: previous ocular trauma, previous ocular surgery, connective tissue disease

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: we plan to enroll 20 consecutive patients with cataract who did not undergo previous surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
cataract lens hardness according to LOCS III classification system | at enrolling
  lens opacity and estimated nucleous hardness according to international LOCS classification
average voltage | at the time of surgery
  voltage necessary to emulsify cataratct nuclous
peak voltage | at the time of surgery
  maximum voltage necessary to emulsify cataract nucleous

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Rossi, MD, Principal Investigator — IRCCS Policlinico San MArtino
Locations (1):
- IRCCS Policlinico San Martino, Genoa, Italy